CLINICAL TRIAL: NCT05129826
Title: The Association Between Periodontal Disease and Malnutrition in a Group of Elderly People in Thailand.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MU-DT/PY-IRB 2019/051.1408
Record Dates: First submitted 2021-09-20; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Periodontal Diseases; Malnutrition
Keywords: periodontal disease; malnutrition; older adult
MeSH Terms: conditions — Periodontal Diseases; Malnutrition

STUDY DESIGN:
Intervention Model Description: Subjects who has aged ≥ 60 years old, not receive periodontal treatment within the previous 6 months, able to read Thai and express verbal communication, functional independent older adults (get ≥ 12 points from Barthel Index for Activities of Daily Living) and cognitive functional independent older adults (get > 23 points from Thai Mental State Examination).
Masking Description: The questionnaire is completed through by the 1st researcher and all clinical data collection will be recorded by the 2nd researcher.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- older adult (Experimental): Subjects who has aged ≥ 60 years old.
  Interventions: Behavioral: the association between periodontitis and malnutrition status

INTERVENTIONS:
Behavioral: the association between periodontitis and malnutrition status — be determine the association between periodontitis and malnutrition status in older adult.

SUMMARY:
This study will be determine the association between periodontitis and malnutrition status in older adult.

DETAILED DESCRIPTION:
Ageing may accompany with an accumulation of diseases and impairments cause by physiological, socioeconomic and psychological changes. The older adults are more prone to nutritional deficiencies due to combination of factors such as ageing, excessive polypharmacy, general health decline, poor socioeconomic status, cognitive decline, poor appetite, impaired efficacy of swallowing and limit eating ability.

Periodontitis is a multifactorial disease predominantly a bacterial infection involving the dental biofilm or dental plaque. Periodontitis increases in extent and severity across a large proportion of the human population with ageing. The effects of ageing on the immune system include distinct alterations in both innate and adaptive immune-cell function and effector biomolecules, resulting in processes reflecting immunosenescence, immunoactivation and inflammaging. Moreover, genetic contribution alters immunity and inflammation that play a role in the dysregulation of host responses in ageing. The combination of chronic antigenic burden and uncontrolled inflammatory response can enhance immunosenescence and ageing-associated disease. Periodontitis also has an effect on food intake, nutritional status and quality of life in older adults.

However the relationship between chronic periodontitis and malnutrition in older adult is not clear and needs further study. In this study will be determine the association between periodontitis and malnutrition status in older adult.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who has aged ≥ 60 years old.
2. Subjects who not receive periodontal treatment within the previous 6 months.
3. Subjects who are able to read Thai and express verbal communication.
4. Subjects who are functional independent older adults (get ≥ 12 points from Barthel Index for Activities of Daily Living) [50, 51].
5. Subjects who are cognitive functional independent older adults (get > 23 points from Thai Mental State Examination) [52].

Exclusion Criteria:

1. Subjects with completely edentulous area.
2. Subjects who require antibiotic prophylaxis for dental examination

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 1 hour
  The nutritional status of the participants will be measured by MNA (Mini Nutritional Assessment) questionnaire. The participants with scores ≥ 24 were classified as having a normal nutritional status, 17 to 23.5 were classified as at risk of malnutrition and <17 were classified as malnutrition.
Periodontal status | 2 hour
  The probing pocket depth and clinical attachment level were collected by clinical data collection. The participants who had 4 or more teeth with 1 or more sites with PPD ≥ 4 mm and with clinical attachment loss ≥ 3 mm at the same site was diagnosed as periodontitis.

SECONDARY OUTCOMES:
Variables that associated with malnutrition in older adult. | 1 month
  The variables that may be associated with malnutrition in all participants were collected. Including, the sociodemographic data and health behavioral information were collected by questionnaires. The anthropometric measurements, masticatory ability, periodontal status, number of teeth and functional tooth units were recorded. The complete data was analyzed for the associated with malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Kanyawat Rattanasuwan, Principal Investigator — Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mahidol University.
Locations (1):
- Kanyawat Rattanasuwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No